CLINICAL TRIAL: NCT04035720
Title: Decision Making in Multiple Sclerosis Care Under Uncertainty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Collaborators: Hoffmann-La Roche (Industry); University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 15-340
Record Dates: First submitted 2019-03-25; First posted 2019-07-29 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Multiple Sclerosis
Keywords: decision making; therapeutic; disease modifying agents; monoclonal antobodies; physicians; neurologists; uncertainty; neuroeconomics
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quantitative risk estimation (Experimental): Participants will be exposed to case-scenarios. Each case scenario provides a description of the current clinical situation (e.g. patient age, current treatment, number of relapses, current EDSS, MRI findings, etc). In addition, participants will see a squared box indicating the probability of risk progression (20%, 25%, 85%, 90%). This information may or may not be accurate to reflect potential errors of risk prediction tools.
  Interventions: Other: Quantitative risk
- Qualitative risk estimation (Active Comparator): Participants will be exposed to the same case-scenarios as the intervention arm. Each case scenario provides a description of the current clinical situation (e.g. patient age, current treatment, number of relapses, current EDSS, MRI findings, etc). In addition, participants will see a squared box indicating a qualitative probability of risk progression (low, high). This information may or may not be accurate to reflect potential errors of risk prediction tools.
  Interventions: Other: Quantitative risk

INTERVENTIONS:
Other: Quantitative risk — Participants will be able to see a square box that represent the estimated risk of disease progression. They will have to elect making a therapeutic decision based on the description of the case-scenario or based on the estimated prediction as represented in the square box.

SUMMARY:
The main objectives of this study are:

i) To determine patient-level, physician-level and health system factors influencing therapeutic decisions in multiple sclerosis (MS) care by applying conjoint discrete experiments.

ii) To determine the prevalence of therapeutic inertia among participating neurologists.

iii) To compare clinical judgement vs. a qualitative or quantitative approach when assessing for a given case-scenario.

iv) To evaluate the influence of decision fatigue in treatment decisions.

DETAILED DESCRIPTION:
The landscape of MS care is changing. Currently, there are over 15 disease modifying agents (DMTs) available to treat MS, with varying availability around the world.

Significant heterogeneity exists in the efficacy and risks associated with these therapies.

Neurologists caring for MS patients face important choices in each medical encounter: 1) continue with the same management, 2) initiate or escalate therapy for a more effective or safer agent, or 3) consider a reassessment within months under the uncertainty of the current status of the patient.

Limited information on how physicians weigh in different factors when making therapeutic decisions.

Physicians (cognitive biases affecting decision making) and health system (e.g. access to an infusion center) factors are the most responsible causes of practice gaps in MS care. The physician's component is the least studied.

Therapeutic inertia (TI) is a common phenomenon in MS care defined as lack of treatment initiation or escalation (e.g. switch interferons or glatiramer to fingolimod /alemtuzumab /natalizumab/ocrelizumab/ etc.) when recommended by guidelines or evidence of disease progression. This phenomenon leads to poorer patient's outcomes, greater disability, and diminished quality of life.

Goals of the study: i) to determine what are the most relevant factors influencing therapeutic decisions among neurologists with expertise in MS care; ii) to asses whether physicians rely on medical information provided in a case scenario versus a quantitative or qualitative estimation of disease progression based on hypothetical models.

ELIGIBILITY:
Inclusion Criteria:

* Actively practicing neurologist
* Expertise in treating patients with multiple sclerosis (at least 12 per year)
* Clinical setting: academic or community institutions, private practice or outpatient clinic
* Certified physicians in their specialty
* Online consent to participate in the study

Ages: 23 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2019-07-06 (Actual); Primary Completion 2021-07-21 (Estimated); Study Completion 2021-12-22 (Estimated)

PRIMARY OUTCOMES:
Therapeutic inertia score | At the completion of the study, an estimated 90 minutes
  The therapeutic inertia (TI) score is based on our previous work published elsewhere (see references). It is based on the sum number of case-scenarios that required treatment escalation over the total number of presented scenarios (10).
  Range: 0 (lowest value) to 10 (maximal value). The higher value represents the higher level of therapeutic inertia. There is no subscale. This measurement has been previously reported (Saposnik et al. JAMA Netw Open. 2019 Jul 3;2(7):e197093. doi: 10.1001/jamanetworkopen.2019.7093; Saposnik et al. MDM Policy Pract. 2019 Jun 21;4(1):2381468319855642. doi: 10.1177/2381468319855642)
Accuracy of treatment decisions | At the completion of the study, an estimated 90 minutes
  Comparison of discordant pairs in each arm: Using chi-square (parametric) test, there will be a comparison between groups (intervention vs. control) in the proportion of participants who made accurate therapeutic decisions.

SECONDARY OUTCOMES:
Therapeutic decisions under fatigue | At the completion of the study, an estimated 90 minutes
  Given that participants will be exposed to several case-scenarios, a comparison of therapeutic inertia will be conducted between the first half and the second half of case scenarios as previously reported (Saposnik et al. Front Neurol. 2017 Aug 21;8:430. doi: 10.3389/fneur.2017.00430. eCollection 2017).
Prevalence of therapeutic inertia (TI) | At the completion of the study, an estimated 90 minutes
  Comparison of treatment decisions using a binary definition of therapeutic inertia (TI). Lack of treatment escalation in at least one case-scenario (out of the total) will be considered as TI present as previously reported ((Saposnik et al. JAMA Netw Open. 2019 Jul 3;2(7):e197093. doi: 10.1001/jamanetworkopen.2019.7093; Saposnik et al. MDM Policy Pract. 2019 Jun 21;4(1):2381468319855642. doi: 10.1177/2381468319855642)
Factors associated with therapeutic decisions | At the completion of the study, an estimated 90 minutes
  Participants will be exposed to 12 pairs of case-scenarios as per the discrete choice design. Participants have to choose the ideal case-scenario (e.g. A, B or neither- but they cannot choose both) for escalating treatment. Each pair of case-scenarios represent a comprehensive combination of possible variables. The most common factors associated with treatment escalation will be assessed based on these experimental design. A weighted estimate will be calculated for each collected variable.
  See details in Discrete Choice Experiment Response Rates: A Meta-analysis.Watson V et al. Health Econ. (2017) and Saposnik et al.Stroke. 2019 Jul 22:STROKEAHA119025631. doi: 10.1161/STROKEAHA.119.025631. [Epub ahead of print]

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Saposnik, MD, MSc, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Saposnik G, Sempere AP, Prefasi D, Selchen D, Ruff CC, Maurino J, Tobler PN. Decision-making in Multiple Sclerosis: The Role of Aversion to Ambiguity for Therapeutic Inertia among Neurologists (DIScUTIR MS). Front Neurol. 2017 Mar 1;8:65. doi: 10.3389/fneur.2017.00065. eCollection 2017. PMID 28298899